CLINICAL TRIAL: NCT06440824
Title: A Multicenter Randomized Controlled Study on the Treatment of Refractory CTIT With Romiplostim N01 Compared to Recombinant Human Thrombopoietin
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-CIT-IIT-001
Record Dates: First submitted 2024-05-23; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: CTIT-Chemotherapy Induced Thrombocytopenia
Keywords: Romiplostim N01，Recombinant Human Thrombopoietin，CTIT
MeSH Terms: interventions — Thrombopoietin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Romiplostim N01 (Experimental)
  Interventions: Drug: Romiplostim N01
- Recombinant Human Thrombopoietin (Active Comparator)
  Interventions: Drug: Recombinant Human Thrombopoietin

INTERVENTIONS:
Drug: Romiplostim N01 — 2.0 µg/kg, subcutaneous injection, once a week, up to a maximum of 8 weeks. Stop medication when platelet count increases by 50 × 109/L or more compared to before medication
  Arms: Romiplostim N01
Drug: Recombinant Human Thrombopoietin — 30000 U/d, subcutaneously injected once a day, for a maximum of 8 weeks. Medication should be stopped when platelets increase by 50 × 109/L or more compared to before medication
  Arms: Recombinant Human Thrombopoietin

SUMMARY:
A Multicenter Randomized Controlled Study on the Treatment of Refractory CTIT With Romiplostim N01 Compared to Recombinant Human Thrombopoietin

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form before enrollment;
2. Age range from 18 to 75 years old;
3. Solid tumors or hematological tumors confirmed by tissue or pathology;
4. CTIT patients caused by anti-tumor therapy;
5. At least 2 weeks of treatment with two types of platelet growth factors and no response (including rhTPO or TPO-RA)
6. Have not received treatment with Roptistine/Roptistine N01;
7. ECOG PS score: 0-2;
8. Platelet value<30 × 109/L;
9. Estimated survival time during screening is ≥ 12 weeks;
10. Subjects of childbearing age agree to take reliable contraceptive measures (including male or female condoms, contraceptive foam, contraceptive gel, contraceptive film, contraceptive cream, contraceptive suppository, abstinence and the placement of intrauterine devices, etc.) throughout the study period; Excluding female participants who have undergone hysterectomy, bilateral salpingectomy, bilateral tubal ligation, or more than 1 year after menopause, as well as male participants who have undergone bilateral salpingectomy or ligation;
11. Voluntarily participate in this study, sign an informed consent form, and have good compliance.

Exclusion Criteria:

-

Patients with any of the following conditions are not eligible for inclusion in this study:

1. Suffering from hematopoietic system diseases other than thrombocytopenia (CIT) caused by tumor chemotherapy drugs, including but not limited to leukemia, primary immune thrombocytopenia, myeloproliferative diseases, multiple myeloma, and myelodysplastic syndrome;
2. Screening for thrombocytopenia caused by causes other than CIT within the first 6 months, including but not limited to chronic liver disease, splenic hyperfunction, infection, and bleeding;
3. Bone marrow invasion or metastasis;
4. Have received pelvic and spinal radiation therapy, as well as bone field radiation therapy, or are currently/expected to receive radiation therapy within the three months prior to screening;
5. Screening for a history of severe cardiovascular disease within the first 6 months, such as congestive heart failure (NYHA heart function score III-IV), known arrhythmias that increase the risk of thromboembolism, such as atrial fibrillation, after coronary stent implantation, angioplasty, and coronary artery bypass grafting;
6. Any history of arterial or venous thrombosis occurring within the first 6 months of screening;
7. Screening for clinical manifestations of severe bleeding within the first two weeks, such as gastrointestinal or central nervous system bleeding;
8. Brain tumors or brain metastases;
9. Urgent treatment is required, such as vena cava syndrome and spinal cord compression syndrome;
10. Neutrophil absolute value < 1.0 × 109/L, hemoglobin < 80g/L, allowing the use of granulocyte colony-stimulating factors and red blood cells that comply with clinical norms EPO infusion therapy;
11. Significant abnormalities in liver function: patients without liver metastasis, ALT/AST>3ULN (upper limit of normal value), TBIL>3ULN； Patients with liver metastasis are present, ALT/AST≥5ULN，TBIL≥5ULN；
12. Renal dysfunction: blood creatinine ≥ 1.5ULN or eGFR ≤ 60 ml/min (Cockcroft Gault formula);
13. Within the first month prior to screening, patients who have received treatment with loperstine/loperstine N01 or recombinant human thrombopoietin (rhTPO);
14. Received platelet transfusion within the first 3 days of randomization;
15. Patients who are known or expected to be allergic or intolerant to Roxetine N01 or rhTPO excipients
16. HIV infected individuals;
17. Pregnant or lactating women;
18. Participated in any clinical study of any other investigational drug or device three months prior to screening;
19. The researchers believe that participating in the trial poses a significant risk to the health or safety of the subjects, or other circumstances that may affect the efficacy evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with PLT ≥ 50 × 109/L within 4 weeks after receiving treatment | Within 4 weeks after receiving treatment

SECONDARY OUTCOMES:
The time required for PLT to recover to 50 × 109/L or above after treatment | up to 8 weeks
The proportion of patients with PLT ≥ 50 × 109/L after 2 weeks of treatment | 2 weeks after receiving treatment
The proportion of patients with PLT ≥ 50 × 109/L after 12 weeks of treatment | 12 weeks after receiving treatment
The lowest platelet count from receiving treatment to the end of treatment | up to 8 weeks
The proportion of patients receiving platelet transfusion | through study completion, an average of 5 months
The proportion of restoring anti-tumor treatment for at least 2 cycles without recurrence of CTIT | through study completion, an average of 5 months